CLINICAL TRIAL: NCT02368145
Title: Inflammation and Post-Stroke Depression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alexander Kusnecov, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Alexander Kusnecov, Ph.D., Professor of Psychology, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 2012001658; pc 62-12 (Other Grant/Funding Number: New Jersey Health Foundation, Inc.)
Record Dates: First submitted 2014-11-04; First posted 2015-02-20 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Stroke; Acute Stroke
Keywords: stroke; acute stroke; post stroke depression
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to see if there is a relationship between stroke, post-stroke depression, and measures of inflammatory and/or stress compounds in the blood. Brain injury, as caused by stroke, leads to an inflammatory response in the brain which in turn can influence inflammatory and stress responses in other parts of the body outside of the brain. These responses can be measured by analyzing various substances in the blood and in the white blood cells. The investigators will measure these substances (cytokines, glucocorticoids) and compare them to the absence, presence, or degree of depression that the investigators will determine by neurological and psychological testing. The investigators will be drawing blood for this study on admission, at or around day 3, at or around day 7 and at or around day 90, which is not part of routine stroke care. The investigators will be asking subjects to participate in answering question/scales on these same days, some of these questionnaires are also not part of routine stroke care. Standard stroke care is being done other than blood drawing/participating in answering questions/scales. Approximately 25 people will be enrolled over one year.

DETAILED DESCRIPTION:
Depression is a common long-term outcome of acute ischemic stroke (AIS), and can impede recovery, increase stroke recurrence, and influence mortality from stroke. Based on literature reviewed below, the investigators propose the novel over-arching hypothesis: that post-stroke depression (PSD) occurs in patients who show elevated production of proinflammatory immune cytokines during and/or after stroke, and at the same time present with reduced sensitivity to the immunosuppressive effects of glucocorticoids, which otherwise would be expected to have down-regulated cytokine production.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be male and female patients with acute ischemic stroke of the brain. Vascular risk factors, including diabetes, hypertension, and coronary artery disease, are expected to be common, and will be recorded in the Source Documents (appendix). Patients will be included if:

  * Aged ≥ 18 years of age
  * Neuroimaging or clinical symptoms are consistent with an acute ischemic stroke (AIS)
  * There are no alternative explanations for symptoms (eg. tumor, witnessed seizure, history of complicated migraine headache, hypoglycemia [blood sugar (BS) < 50 mg/dL] or hyperglycemia (BS > 400 mg/dL)
  * Subject is able to be enrolled and have blood samples drawn (Note: inability to provide a sample within 48 hours does not preclude inclusion if consent is provided after this time and patient can provide blood at subsequent time points (see Table)
  * Subject is able to provide informed consent for participation in this research study

Exclusion Criteria:

* • Other known severe/terminal illness which limits life expectancy to < 90 days, sepsis, disseminated intravascular coagulopathy (DIC), infective endocarditis, metastatic cancer, or cerebral vasculitis

  * Current diagnosis of or treatment for major depressive disorder
  * Women who are pregnant at the time of stroke, since pregnancy alters inflammatory markers
  * Communication problems due to aphasia at visit 2, inability to speak English
  * History of substance abuse and other relevant psychiatric conditions
  * Autoimmune, current or recent infection, hematological disorders, use of immune modulating drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with acute iechemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
• The analysis of the presence of specific inflammatory markers | 90 days
  • Analysis of blood for the presence of Increased proinflammatory cytokines measured in blood plasma and isolated peripheral blood mononuclear cells (PBMC),reduced sensitivity to the suppressive effects of the synthetic glucocorticoid, dexamethasone, on cytokine production and proliferation in stimulated PBMC cultures and high cortisol and ACTH levels
presence of depression in people with ischemic stroke | 90 days
  Continuous measures of clinician-rated depression severity and potential co-morbid anxiety will be measured with the Hamilton Depression and Anxiety Scales (Ham-A and Ham-D 46-48). These are widely-used and well-validated rating scales that have been used in a variety of patient populations, and will be supplemented for thoroughness with the Beck Depression Inventory. The presence and history of depression and anxiety disorders will be also be assessed using the Structured Diagnostic Interview for Axis I DSM-IV Disorders depression and anxiety modules (SCID) 49. The SCID is a diagnostic semi-structured interview designed to assess and diagnose mental illnesses as defined by the DSM-IV (American Psychiatric Association, 2000), which is the gold standard for diagnosis categorization in the United States.

SECONDARY OUTCOMES:
Measurement and identification stroke location | 90 days
  Localization will occur through neuroimaging by either CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: James S McKinney, MD, Principal Investigator — Rutgers University; Alexander Kusnecov, PhD, Study Director — Rutgers University
Locations (1):
- Rutgers, The State University, New Brunswick, New Jersey, United States